CLINICAL TRIAL: NCT07142226
Title: Role of Circulating Tumor DNA (ctDNA) in Genetic Profiling and Clinical Outcomes for Advanced Biliary Tract Cancer (BTC) Patients - A Multicenter, Prospective, Observational Epidemiology Study
Brief Title: Role of ctDNA in Genetic Profiling & Outcomes for Advanced BTC
Status: Not yet recruiting | Type: Observational
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Hong Jae Chon, Principal Investigator, CHA University
Other Study IDs: CHAMC2025-03-043
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary Tract Cancer; Biomarker; IDH1 mutation; FGFR2 fusion; Biomarker Analysis; Circulating Tumor DNA (ctDNA)
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Circulating Tumor DNA; Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Advanced BTC Patients: Description: Patients with histologically or cytologically confirmed advanced biliary tract cancer (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer) who are enrolled prospectively across participating centers in Korea.
  Number of Participants: 200 (anticipated)
  Cohort Type: Single observational cohort
  Interventions: Genetic: Circulating Tumor DNA (ctDNA) Testing (ctDNA-based Next-Generation Sequencing (NGS))

INTERVENTIONS:
Genetic: Circulating Tumor DNA (ctDNA) Testing (ctDNA-based Next-Generation Sequencing (NGS)) — Peripheral blood will be collected from patients with advanced biliary tract cancer for circulating tumor DNA (ctDNA) testing. Next-generation sequencing (NGS) will be performed to detect clinically relevant genomic alterations, including IDH1 mutations, FGFR2 fusions, ERBB2 amplifications, and MSI-H/dMMR. The ctDNA results will be compared with tissue-based genomic profiling to evaluate concordance and clinical utility.
  Other Names: Liquid Biopsy, Alpha Liquid 100

SUMMARY:
Biliary tract cancer (BTC) is a rare and heterogeneous disease with high incidence and mortality in Korea. Molecular profiling has enabled the identification of actionable alterations such as Isocitrate Dehydrogenase 1 (IDH1) mutations, FGFR2 fusions, ERBB2 amplifications, and dMMR/MSI-H status. However, the utility of tumor tissue-based next-generation sequencing (NGS) is often limited by difficulties in obtaining adequate tissue samples and the lack of in-house sequencing capacity across many hospitals.

Circulating tumor DNA (ctDNA) analysis offers a minimally invasive alternative that can provide rapid and reliable genomic profiling. In a previous study, ctDNA testing showed high concordance with tissue-based genomic profiling for clinically significant alterations, particularly IDH1 mutations, and identified additional mutations not detected in tumor tissue. These findings suggest that ctDNA may expand access to targeted therapies such as ivosidenib .

This multicenter, prospective, observational epidemiology study, organized by the Korean Cancer Study Group (KCSG) Biliary Tract Cancer Subcommittee, will evaluate the clinical utility of ctDNA-based genomic profiling in patients with advanced BTC. The study will assess concordance between ctDNA and tumor tissue sequencing, describe the prevalence of actionable alterations, and explore the impact of ctDNA testing on treatment decisions and clinical outcomes. By leveraging a nationwide network of BTC specialists, this study seeks to validate ctDNA as a feasible and scalable tool for precision oncology, supporting timely and personalized therapy for patients with BTC.

DETAILED DESCRIPTION:
Biliary tract cancer (BTC) encompasses a rare and diverse group of tumors characterized by varying anatomical locations-including extrahepatic, intrahepatic, and gallbladder lesions. Therapeutic innovations in advanced BTC are hindered by the rarity and heterogeneity of its subtypes, with particularly high incidence and mortality rates observed in Korea.

Recent advances in molecular profiling have enabled the identification of potential therapeutic targets for BTC. These findings have led to the approval of several therapies for BTC, including those targeting IDH1 mutations, FGFR2 fusions, ERBB2 amplifications, as well as immunotherapies for DNA mismatch repair-deficient (dMMR) or microsatellite instability-high (MSI-H) subtypes. Genomic profiling is essential to detect these targetable alterations, helping to guide appropriate, targeted therapies for patients with BTC. Traditional genomic profiling is typically conducted using formalin-fixed paraffin-embedded (FFPE) tumor tissues; therefore, the challenge of obtaining adequate tumor tissue samples in BTC can impede molecular evaluations. Circulating tumor DNA (ctDNA) from blood may offer an alternative to tissue-based analysis.

In a previous study, the investigators assessed the concordance between ctDNA and tissue genomic profiling in a large cohort of Asian patients with advanced BTC and evaluated the feasibility of liquid biopsy in the treatment of BTC. As a result, ctDNA-based genotyping exhibited acceptable concordance with tissue genomic profiling for clinically significant mutations classified as tier 1 or 2, with a sensitivity of 84.8% and a positive predictive value (PPV) of 79.4%. Notably, high concordance of actionable alterations between ctDNA and tissue for IDH1 mutations was observed, with 100% sensitivity (5/5) and 71.4% PPV (5/7), and for FGFR2 fusions with 66.7% sensitivity (2/3) and 100% PPV (2/2). Additionally, using ctDNA, five IDH1 mutations were identified in tissue samples and two additional IDH1 mutations were detected only in ctDNA.

The IDH1 mutations have significant clinical implications for patients with BTC due to their considerable frequency (approximately 13% in intrahepatic cholangiocarcinoma; range, 9-20%) and the availability of targeted therapy; ivosidenib was approved by both the U.S. Food and Drug Administration (FDA) and the Ministry of Food and Drug Safety (MFDS) in Korea. Although relatively high concordance between ctDNA and tumor tissue for IDH1 mutations was found, the occurrence of these alterations was low, and a more comprehensive comparative analysis is warranted. Therefore, the validation of ctDNA genomic profiling in a larger cohort of patients with BTC is not just a suggestion, but a pressing need to establish its potential as a promising approach for guiding personalized treatment strategies.

Justification for ctDNA in BTC:

The Korean Cancer Study Group (KCSG) Biliary Tract Cancer Subcommittee includes nearly 100 specialists from hospitals across the country. However, not all hospitals in Korea have in-house capabilities for NGS (Next-Generation Sequencing), making it challenging to implement NGS as recommended in biliary tract cancer treatment guidelines. In contrast, ctDNA allows for the detection of a patient's genetic alterations through a simple, non-invasive blood sampling process. This method can identify targetable alterations, facilitating appropriate treatments. Additionally, ctDNA offers a shorter turnaround time, which can help shorten diagnostic timelines and streamline patient access to treatments like ivosidenib.

Long-Term Benefits:

As demonstrated in a recently published study by Immune & Biotech Diagnostics (IMBDx, Seoul, South Korea), IMBDx's ctDNA test, Alpha Liquid 100, not only identified all five cases of IDH1 mutation detected by conventional tissue NGS but also identified two additional IDH1 mutations that tissue NGS failed to detect. This capability could enable more patients to access treatment with ivosidenib. Moreover, if ctDNA-based NGS testing becomes routine within the KCSG Biliary Tract Cancer Subcommittee, which includes a substantial number of specialists dedicated to treating biliary tract cancer in Korea, it is likely that the use of ctDNA for IDH1 mutation detection will continue beyond this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed advanced or metastatic biliary tract cancer (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer).
* Patients who meet one of the following conditions:

  * Patients prior to initiation of first-line systemic chemotherapy, or
  * Patients previously treated with systemic chemotherapy who can provide a blood sample immediately before starting subsequent therapy.
* Age ≥ 19 years at the time of enrollment.
* Willingness to provide a blood sample for ctDNA analysis.

Exclusion Criteria:

* Patients who refuse to provide blood samples for ctDNA testing.
* Patients unable to provide written informed consent.
* Patients concurrently enrolled in a similar study within the same institution. Prior screening will be performed to prevent duplicate enrollment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed advanced or metastatic biliary tract cancer, including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer. Eligible patients are either treatment-naïve prior to first-line systemic chemotherapy or previously treated patients able to provide a blood sample before starting subsequent therapy. All participants must be 19 years of age or older and willing to provide blood samples for ctDNA analysis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Concordance Between ctDNA and Tissue-Based Genomic Profiling | Within 4 weeks of study enrollment, prior to initiation of systemic therapy
  The proportion of concordance between circulating tumor DNA (ctDNA)-based next-generation sequencing (NGS) and tissue-based genomic profiling in detecting clinically relevant genetic alterations (e.g., IDH1 mutations, FGFR2 fusions, ERBB2 amplifications, MSI-H/dMMR) among patients with advanced biliary tract cancer.

SECONDARY OUTCOMES:
Detection Rate of Actionable Alterations using ctDNA | At baseline (prior to treatment initiation, within 4 weeks of enrollment)
  To determine the detection rate of clinically significant alterations such as IDH1 mutations, FGFR2 fusions, and ERBB2 amplifications by ctDNA analysis.
Positive Predictive Value (PPV) and Sensitivity of ctDNA | At baseline (prior to treatment initiation, within 4 weeks of enrollment)
  To assess the PPV and sensitivity of ctDNA profiling compared with matched tissue NGS results.
Feasibility of ctDNA Testing in Clinical Practice | From baseline through study completion, up to 24 months
  To evaluate the feasibility of ctDNA analysis in a real-world multicenter setting, including sample collection success rate, assay success rate, and turnaround time.

OTHER OUTCOMES:
Correlation between Genetic Alterations and Clinical Outcomes | From baseline through follow-up, up to 36 months
  To explore associations between specific genetic alterations (e.g., IDH1 mutations, FGFR2 fusions) and clinical outcomes such as overall survival (OS), progression-free survival (PFS), and objective response rate (ORR).
Identification of ctDNA-only Mutations | At baseline (prior to treatment initiation, within 4 weeks of enrollment)
  To investigate genetic alterations detected exclusively by ctDNA but not by tissue-based NGS, with a particular focus on IDH1 mutations.
Implementation within KCSG Biliary Tract Cancer Network | From baseline through study completion, up to 24 months
  To assess the potential for ctDNA-based genomic testing to be integrated into routine practice across the Korean Cancer Study Group (KCSG) Biliary Tract Cancer Subcommittee network and its implications for future treatment guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jae Chon, MD. PhD, Principal Investigator — Principal Investigator
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baria K, De Toni EN, Yu B, Jiang Z, Kabadi SM, Malvezzi M. Worldwide Incidence and Mortality of Biliary Tract Cancer. Gastro Hep Adv. 2022 Apr 15;1(4):618-626. doi: 10.1016/j.gastha.2022.04.007. eCollection 2022. PMID 39132071
- [Background] Valle JW, Lamarca A, Goyal L, Barriuso J, Zhu AX. New Horizons for Precision Medicine in Biliary Tract Cancers. Cancer Discov. 2017 Sep;7(9):943-962. doi: 10.1158/2159-8290.CD-17-0245. Epub 2017 Aug 17. PMID 28818953
- [Background] Abou-Alfa GK, Macarulla T, Javle MM, Kelley RK, Lubner SJ, Adeva J, Cleary JM, Catenacci DV, Borad MJ, Bridgewater J, Harris WP, Murphy AG, Oh DY, Whisenant J, Lowery MA, Goyal L, Shroff RT, El-Khoueiry AB, Fan B, Wu B, Chamberlain CX, Jiang L, Gliser C, Pandya SS, Valle JW, Zhu AX. Ivosidenib in IDH1-mutant, chemotherapy-refractory cholangiocarcinoma (ClarIDHy): a multicentre, randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Jun;21(6):796-807. doi: 10.1016/S1470-2045(20)30157-1. Epub 2020 May 13. PMID 32416072
- [Background] Zhu AX, Macarulla T, Javle MM, Kelley RK, Lubner SJ, Adeva J, Cleary JM, Catenacci DVT, Borad MJ, Bridgewater JA, Harris WP, Murphy AG, Oh DY, Whisenant JR, Lowery MA, Goyal L, Shroff RT, El-Khoueiry AB, Chamberlain CX, Aguado-Fraile E, Choe S, Wu B, Liu H, Gliser C, Pandya SS, Valle JW, Abou-Alfa GK. Final Overall Survival Efficacy Results of Ivosidenib for Patients With Advanced Cholangiocarcinoma With IDH1 Mutation: The Phase 3 Randomized Clinical ClarIDHy Trial. JAMA Oncol. 2021 Nov 1;7(11):1669-1677. doi: 10.1001/jamaoncol.2021.3836. PMID 34554208
- [Background] Abou-Alfa GK, Sahai V, Hollebecque A, Vaccaro G, Melisi D, Al-Rajabi R, Paulson AS, Borad MJ, Gallinson D, Murphy AG, Oh DY, Dotan E, Catenacci DV, Van Cutsem E, Ji T, Lihou CF, Zhen H, Feliz L, Vogel A. Pemigatinib for previously treated, locally advanced or metastatic cholangiocarcinoma: a multicentre, open-label, phase 2 study. Lancet Oncol. 2020 May;21(5):671-684. doi: 10.1016/S1470-2045(20)30109-1. Epub 2020 Mar 20. PMID 32203698
- [Background] Javle M, Roychowdhury S, Kelley RK, Sadeghi S, Macarulla T, Weiss KH, Waldschmidt DT, Goyal L, Borbath I, El-Khoueiry A, Borad MJ, Yong WP, Philip PA, Bitzer M, Tanasanvimon S, Li A, Pande A, Soifer HS, Shepherd SP, Moran S, Zhu AX, Bekaii-Saab TS, Abou-Alfa GK. Infigratinib (BGJ398) in previously treated patients with advanced or metastatic cholangiocarcinoma with FGFR2 fusions or rearrangements: mature results from a multicentre, open-label, single-arm, phase 2 study. Lancet Gastroenterol Hepatol. 2021 Oct;6(10):803-815. doi: 10.1016/S2468-1253(21)00196-5. Epub 2021 Aug 3. PMID 34358484
- [Background] Javle M, Borad MJ, Azad NS, Kurzrock R, Abou-Alfa GK, George B, Hainsworth J, Meric-Bernstam F, Swanton C, Sweeney CJ, Friedman CF, Bose R, Spigel DR, Wang Y, Levy J, Schulze K, Cuchelkar V, Patel A, Burris H. Pertuzumab and trastuzumab for HER2-positive, metastatic biliary tract cancer (MyPathway): a multicentre, open-label, phase 2a, multiple basket study. Lancet Oncol. 2021 Sep;22(9):1290-1300. doi: 10.1016/S1470-2045(21)00336-3. Epub 2021 Jul 30. PMID 34339623
- [Background] Le DT, Kim TW, Van Cutsem E, Geva R, Jager D, Hara H, Burge M, O'Neil B, Kavan P, Yoshino T, Guimbaud R, Taniguchi H, Elez E, Al-Batran SE, Boland PM, Crocenzi T, Atreya CE, Cui Y, Dai T, Marinello P, Diaz LA Jr, Andre T. Phase II Open-Label Study of Pembrolizumab in Treatment-Refractory, Microsatellite Instability-High/Mismatch Repair-Deficient Metastatic Colorectal Cancer: KEYNOTE-164. J Clin Oncol. 2020 Jan 1;38(1):11-19. doi: 10.1200/JCO.19.02107. Epub 2019 Nov 14. PMID 31725351
- [Background] Lamarca A, Kapacee Z, Breeze M, Bell C, Belcher D, Staiger H, Taylor C, McNamara MG, Hubner RA, Valle JW. Molecular Profiling in Daily Clinical Practice: Practicalities in Advanced Cholangiocarcinoma and Other Biliary Tract Cancers. J Clin Med. 2020 Sep 3;9(9):2854. doi: 10.3390/jcm9092854. PMID 32899345
- [Background] Strickler JH, Loree JM, Ahronian LG, Parikh AR, Niedzwiecki D, Pereira AAL, McKinney M, Korn WM, Atreya CE, Banks KC, Nagy RJ, Meric-Bernstam F, Lanman RB, Talasaz A, Tsigelny IF, Corcoran RB, Kopetz S. Genomic Landscape of Cell-Free DNA in Patients with Colorectal Cancer. Cancer Discov. 2018 Feb;8(2):164-173. doi: 10.1158/2159-8290.CD-17-1009. Epub 2017 Dec 1. PMID 29196463
- [Background] Goyal L, Saha SK, Liu LY, Siravegna G, Leshchiner I, Ahronian LG, Lennerz JK, Vu P, Deshpande V, Kambadakone A, Mussolin B, Reyes S, Henderson L, Sun JE, Van Seventer EE, Gurski JM Jr, Baltschukat S, Schacher-Engstler B, Barys L, Stamm C, Furet P, Ryan DP, Stone JR, Iafrate AJ, Getz G, Porta DG, Tiedt R, Bardelli A, Juric D, Corcoran RB, Bardeesy N, Zhu AX. Polyclonal Secondary FGFR2 Mutations Drive Acquired Resistance to FGFR Inhibition in Patients with FGFR2 Fusion-Positive Cholangiocarcinoma. Cancer Discov. 2017 Mar;7(3):252-263. doi: 10.1158/2159-8290.CD-16-1000. Epub 2016 Dec 29. PMID 28034880
- [Background] Miller AM, Shah RH, Pentsova EI, Pourmaleki M, Briggs S, Distefano N, Zheng Y, Skakodub A, Mehta SA, Campos C, Hsieh WY, Selcuklu SD, Ling L, Meng F, Jing X, Samoila A, Bale TA, Tsui DWY, Grommes C, Viale A, Souweidane MM, Tabar V, Brennan CW, Reiner AS, Rosenblum M, Panageas KS, DeAngelis LM, Young RJ, Berger MF, Mellinghoff IK. Tracking tumour evolution in glioma through liquid biopsies of cerebrospinal fluid. Nature. 2019 Jan;565(7741):654-658. doi: 10.1038/s41586-019-0882-3. Epub 2019 Jan 23. PMID 30675060
- [Background] Hwang S, Woo S, Kang B, Kang H, Kim JS, Lee SH, Kwon CI, Kyung DS, Kim HP, Kim G, Kim C, Chon HJ. Concordance of ctDNA and tissue genomic profiling in advanced biliary tract cancer. J Hepatol. 2025 Apr;82(4):649-657. doi: 10.1016/j.jhep.2024.10.020. Epub 2024 Oct 21. PMID 39442892
- [Background] Boscoe AN, Rolland C, Kelley RK. Frequency and prognostic significance of isocitrate dehydrogenase 1 mutations in cholangiocarcinoma: a systematic literature review. J Gastrointest Oncol. 2019 Aug;10(4):751-765. doi: 10.21037/jgo.2019.03.10. PMID 31392056